CLINICAL TRIAL: NCT00003288
Title: A Trial of Tirapazamine and Cyclophosphamide in Children With Refractory Solid Tumors
Brief Title: Tirapazamine Plus Cyclophosphamide in Treating Children With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01837; POG-9675; CDR0000066219 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2000-04

CONDITIONS: Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — Filgrastim; Cyclophosphamide; Tirapazamine

ARMS (1):
- Arm I (Experimental): See arm description.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: tirapazamine

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: tirapazamine

SUMMARY:
Phase I trial to study the effectiveness of tirapazamine plus cyclophosphamide in treating children who have refractory solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose and the dose limiting toxicity of tirapazamine when administered with cyclophosphamide as intravenous infusions to children with refractory solid tumors.

II. Determine the incidence and severity of other toxicities of tirapazamine and cyclophosphamide in these patients.

III. Determine a safe and tolerable dose of tirapazamine administered with cyclophosphamide for a phase II study for the same indications.

IV. Determine the pharmacokinetics of tirapazamine in children and adolescents receiving the combination of tirapazamine and cyclophosphamide.

V. Determine the preliminary evidence of antitumor activity of tirapazamine and cyclophosphamide.

OUTLINE: This is a dose escalation study.

Patients receive tirapazamine by 2 hour intravenous infusion (hours 0-2) followed 2 hours later by a 30 minute intravenous infusion of cyclophosphamide. This course is repeated every 3 weeks in patients with partial/complete response or stable disease for a maximum of 1 year. Cohorts of 3-6 patients each are treated at each dose level of tirapazamine. Dose escalation of tirapazamine occurs when 0 of 3 patients or 1 of 6 patients has experienced dose limiting toxicity (DLT). If DLT is experienced in 1 of 3 patients at a given dose level, up to 3 additional patients are treated at that same dose level. If none of the 3 additional patients at that dose level experiences DLT, the dose is escalated. If DLT is experienced in 1 or more of the additional 3 patients, the maximum tolerated dose (MTD) has been exceeded and 3 patients are treated at the next lower dose level (defined as the MTD). A total of six patients are treated at the MTD. If DLT is proved to be neutropenia, patients must then also meet the additional eligibility criteria listed for stratum 2. If neutropenia continues to be the DLT in stratum 2, then additional patients receive subcutaneous filgrastim (granulocyte colony-stimulating factor; G-CSF) beginning 24 hours after cyclophosphamide. A second MTD may be determined for chemotherapy with G-CSF. Patients are followed every 6 months for 4 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor that is refractory to conventional therapy or for which no effective therapy is known
* Brain tumors eligible Brainstem gliomas may waive histological verification requirement
* Neurologic deficits associated with CNS malignancies must be stable for a minimum of 4 weeks prior to study
* No leukemia Stratum 2
* No marrow involvement

PATIENT CHARACTERISTICS:

* Age: 21 and under
* Performance status: Karnofsky or Lansky 50-100%
* Life expectancy: At least 8 weeks
* Absolute neutrophil count at least 1,000/mm3
* Platelet count at least 75,000/mm3
* Hemoglobin at least 9 g/dL
* Bilirubin less than 1.5 mg/dL
* SGPT less than 5 times normal
* Creatinine normal for age OR creatinine clearance at least 70 mL/min
* Shortening fraction at least 27% of normal OR ejection fraction greater than 50% of normal
* Not pregnant or nursing
* Negative pregnancy test required

PRIOR CONCURRENT THERAPY:

* No concurrent anticancer therapy
* At least 6 months since bone marrow transplant and no evidence of graft versus host disease
* At least 1 week since growth factors
* No concurrent granulocyte colony-stimulating factor
* Recovered from prior immunotherapy
* Stratum 2: No prior bone marrow transplantation (with or without total body irradiation)
* At least 6 weeks since prior nitrosourea
* At least 2 weeks since other prior myelosuppressive chemotherapy
* Dexamethasone must be a stable or decreasing dose for 2 weeks prior to study
* Recovered from prior chemotherapy
* Stratum 2: No more than 2 prior chemotherapy regimens
* At least 2 weeks since local palliative radiotherapy (small port)
* At least 6 months since prior substantial bone marrow radiation (e.g., cross- sectional radiotherapy [greater than 24 Gy], total body irradiation, hemi- pelvic radiotherapy)
* Recovered from prior radiotherapy
* Stratum 2: No prior central axis radiation

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 1998-08; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Aquino, MD, Study Chair — Simmons Cancer Center
Locations (28):
- United States (25):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California San Diego Cancer Center, La Jolla, California
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec